CLINICAL TRIAL: NCT00718198
Title: Effects of a Computerized Physician Order Entry (CPOE)-Based Inpatient Insulin Protocol on Glycemic Outcomes
Status: Completed | Type: Observational
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Yannis Guerra, MD, Cook County Health
Other Study IDs: 06-063 JHSEndo01
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
Keywords: Inpatient; Computer Physician Order Entry; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-protocol group: Group admitted 1 (one) month before CPOE protocol changes were made
- Post-protocol group: Group admitted 1 (one) year after CPOE protocol changes were made

SUMMARY:
Retrospective cross-sectional study measuring the impact of a computer=based insulin correction protocol and nursing inservicing on diabetes outcomes

DETAILED DESCRIPTION:
This study is a retrospective cross-sectional study at one institution, where the investigators compared diabetic patients admitted to Medicine Services from March-April 2006 (before CPOE was implemented) to patients admitted from October-November 2007 (one year after CPOE implementation). Capillary blood glucose values, Hemoglobin AIC, diabetes medication profile and demographic data were obtained to compare between groups. The investigators hypothesized that a computer-based protocol that emphasizes basal-bolus and correctional insulin orders and excludes sliding scale, in conjunction with nursing personnel inservicing, improves outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetes Mellitus

Exclusion Criteria:

* Admitted to Non-Medicine Hospital Services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients admitted to Medicine Services
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean Inpatient Glucose | From day of admission to hospital until day of discharge from hospital
  Baseline glucose

SECONDARY OUTCOMES:
Percentage of normoglycemic (70 to 150 mg/dl) patient-days | From day of admission to hospital until day of discharge from hospital
  Percentage of inpatient days at glucose target
Percentage of hyperglycemic patient-days | From day of admission to hospital until day of discharge from hospital
  Percentage of inpatient days above glucose target
Percentage of Patient-days with glucose less than 70 mg/dl | From day of admission to hospital until day of discharge from hospital
  Percentage of inpatient days below glucose target
Percentage of Patients with inpatient or recent (less than 6 months) hemoglobin AIC | From day of admission to hospital until day of discharge from hospital
  Percentage of patients with recent A1c
Length of stay | From day of admission to hospital until day of discharge from hospital
  Number of days inpatient
Distribution of oral hypoglycemic use | From day of admission to hospital until day of discharge from hospital
  Rate of oral diabetes medication use
Distribution of type of insulin therapy used | From day of admission to hospital until day of discharge from hospital
  Rate of insulin use
Percent of patient-days with severe hypoglycemia | From day of admission to hospital until day of discharge from hospital
  Percentage of patient days with glucose below 55 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Yannis S Guerra, MD, Principal Investigator — Rush University Hospital/John H Stroger Jr. Hospital; Krishna Das, MD, Study Chair — John H. Stroger Jr. Hospital; Pete Antonopoulos, MD, Study Chair — John H. Stroger Jr. Hospital; Irene Benson, RN, Study Chair — John H. Stroger Jr. Hospital; Shane Borkowski, MD, Study Chair — John H. Stroger Jr. Hospital; Leon Fogelfeld, MD, Study Chair — John H. Stroger Jr. Hospital; Melanie Gordon, MD, Study Chair — John H. Stroger Jr. Hospital; Betsy Palal, MD, Study Chair — John H. Stroger Jr. Hospital; Joana Witsil, MD, Study Chair — John H. Stroger Jr. Hospital; Evelyn Lacuesta, MD, Study Director — John H. Stroger Jr. Hospital
Locations (1):
- John H. Stroger Jr. Hospital, Chicago, Illinois, United States